CLINICAL TRIAL: NCT02393495
Title: A Further Step Towards Painless Intrauterine Device Insertion, a Randomized Control Trial
Brief Title: Ultrasound Guided Intra-uterine Device Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Dina Mohamed Refaat Dakhly, Lecturer of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22012015
Record Dates: First submitted 2015-01-23; First posted 2015-03-19 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound guided group (Experimental): the female will be asked to be full bladder. the trans-abdominal probe will be placed by an assistant on the suprapubic region. under speculum examination, the intrauterine device IUD (TCu 380A) will be placed till it reaches the fundus of the uterus and then released.
  Interventions: Device: intrauterine device TCu 380A
- Non ultrasound guided group (Experimental): the intrauterine device TCu 380A will be inserted in the conventional method, and checked afterwards by transvaginal ultrasound.
  Interventions: Device: intrauterine device TCu 380A

INTERVENTIONS:
Device: intrauterine device TCu 380A
  Other Names: TCu 380A

SUMMARY:
Different studies have been made in an attempt to reduce the pain and the duration of the process of outpatient insertion of the intrauterine device. in this trial, the investigators aim to insert the IUD under ultrasonographic guidance, which can help to reduce the pain, decrease the process of insertion, in addition, it reduces the incidence of malposition of IUD as well as the risk of complications.

ELIGIBILITY:
Inclusion Criteria:

* Females desiring contraception with the use of IUD

Exclusion Criteria:

* Are pregnant or think they may be pregnant
* Septic pregnancy or abortion
* Have unexplained abnormal vaginal bleeding
* Have untreated cervical cancer
* Have malignant gestational trophoblastic disease
* Have uterine cancer
* Have uterine abnormalities
* Have or may have had a pelvic infection within the past three months
* Have or may have any sexually transmitted disease
* Have pelvic tuberculosis
* Are postpartum between 48 hours and 4 weeks
* Have benign gestational trophoblastic disease
* Have ovarian cancer
* Have AIDS (unless clinically well on anti-retroviral therapy)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Assessment of degree of pain during IUD insertion | 6 months
  Pain will be assessed by the use of visual analog scale, Pain rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Dina MR Dakhly, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr el ainy hospital, Cairo, Egypt